CLINICAL TRIAL: NCT01843985
Title: Observational Study of Survival Times of Stage IV Cancer Patients
Brief Title: Observational Study of Survival Outcomes of Stage IV Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cure Cancer Worldwide Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: YLDZH-OS-1
Record Dates: First submitted 2013-04-27; First posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Stage IV Cancer (Solid Tumors Only); Survival
Keywords: Stage IV cancer; Survival
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1. Eligible RCT/Elect RCT: Eligible for regular chemotherapy, elects and receives regular chemotherapy
- 2. Eligible RCT/Elect LDC: Eligible for regular chemotherapy, elects and receives low-dose chemotherapy
- 3. Eligible RCT/Elect PCO: Eligible for regular chemotherapy, elects and receives palliative care only
- 4. Ineligible RCT/Elect LDC: Ineligible for regular chemotherapy, elects and receives low-dose chemotherapy
- 5. Ineligible RCT/Elect PCO: Ineligible for regular chemotherapy, elects and receives palliative care only

SUMMARY:
Patients diagnosed with Stage IV cancer (solid tumors only) are evaluated to determine whether they are candidates for traditional chemotherapy. If eligible, patients are offered traditional chemotherapy, low-dose chemotherapy, or palliative care. If ineligible, patients are offered low-dose chemotherapy or palliative care. Patients will be monitored for 5 years and survival data recorded.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with Stage IV cancer (solid tumors only)

Exclusion Criteria:

* Patient declines inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
survival | months 1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 60

CONTACTS AND LOCATIONS:
Locations (1):
- Yang Ling Demonstration Zone Hospital, Yangling, Shaanxi, China